CLINICAL TRIAL: NCT07163520
Title: Shear-Wave Elastography Evaluation of the Gastrocnemius Muscle in Children With Idiopathic Toe Walking Compared to Typically Developing Peers
Brief Title: Elastographic Assessment of Gastrocnemius Muscle Structure in Children With Idiopathic Toe Walking
Status: Completed | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Sude Gözüküçük Türkyılmaz, Medical Doctor, Fatih Sultan Mehmet Training and Research Hospital
Other Study IDs: ITW-SWE
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Idiopathic Toe-walking
Keywords: idiopathic toe-walking; shear wave elastography; gastrocnemius; achilles

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Idiopathic Toe Walking Group: Children aged 4 to 12 years with bilateral idiopathic toe-walking pattern, defined as toe-walking gait in the absence of any underlying neurological, orthopedic, or psychiatric conditions (such as cerebral palsy, muscular dystrophies, neuropathies, autism spectrum disorder, or developmental delay).
- Healthy Control Group: Age- and sex-matched typically developing children without a history of toe-walking or any neurological, orthopedic, or psychiatric disorders.

SUMMARY:
Idiopathic toe walking (ITW) is a gait pattern characterized by the absence of heel strike during the stance phase and incomplete foot contact with the ground. After excluding neurological, neuromuscular, and orthopedic causes such as cerebral palsy, neuropathies, myopathies, and spinal dysraphism, the diagnosis of ITW can be established. Although alterations in muscle histology and architecture have been reported in children with ITW, radiological evaluation of the musculoskeletal system remains limited.

Shear Wave Elastography (SWE) is a non-invasive, objective, and cost-effective imaging technique that quantitatively assesses tissue stiffness by measuring shear wave velocity and elasticity.

The present study aims to evaluate gastrocnemius muscle and Achilles tendon elasticity in children with ITW compared with age-matched healthy controls. By combining SWE measurements with clinical assessments-including ankle dorsiflexion range of motion, Toe Walking Severity Scale, Foot Posture Index, and a functionality questionnaire-we aim to better characterize the musculoskeletal alterations associated with ITW.

DETAILED DESCRIPTION:
In some children, the inability to perform heel strike may lead to toe walking. Toe walking can occur due to a variety of conditions, including cerebral palsy, spina bifida, muscular dystrophies, limb-length discrepancies, and autism spectrum disorders. When no underlying medical cause is identified, the diagnosis of idiopathic toe walking (ITW) is made. ITW is a diagnosis of exclusion.

The etiology of ITW remains unclear. A positive family history of toe walking has been frequently reported, suggesting a potential genetic component. Sensory integration deficits have also been proposed as a contributing factor. Muscle biopsy studies have shown an increased proportion of type I fibers in children with ITW compared to typically developing peers. Toe walking leads to remodeling of the muscle-tendon unit. A study using ultrasonography (US), isokinetic dynamometry, and surface electromyography have demonstrated that the gastrocnemius (GC) muscle and its fascicles are longer and the Achilles tendon is shorter in children with ITW compared to healthy controls.

Rehabilitation strategies such as stretching, strengthening, and spasticity management aim to improve the biomechanical properties of the muscle. Investigating biomechanical characteristics, including muscle stiffness, is essential for understanding musculoskeletal adaptations.

Non-invasive techniques are particularly preferred in the pediatric population. Shear-Wave Elastography (SWE) is a non-invasive, cost-effective, and objective method for evaluating tissue stiffness in vivo, with promising clinical applications in the musculoskeletal system. While SWE has been applied in pediatric neuromuscular conditions, data on musculoskeletal imaging in children with ITW remain limited. Few studies have evaluated this population using ultrasonography and none have directly compared ITW children with healthy controls using SWE.

Evaluating differences between children with ITW and their typically developing peers may enhance understanding of this poorly understood gait pattern and support the development of more effective treatment approaches. The aim of this study is to assess the structure of the medial gastrocnemius muscle and Achilles tendon in children with ITW using SWE, comparing the results with a healthy control group. This approach will allow comprehensive evaluation of clinical parameters and musculoskeletal characteristics in this children.

ELIGIBILITY:
Inclusion Criteria:

Children aged 4 to 12 years with a bilateral idiopathic toe walking pattern Absence of neurological, orthopedic, or psychiatric conditions that could explain the toe walking gait pattern (e.g., cerebral palsy, myopathies, autism spectrum disorders, developmental disorders, neuropathies) Healthy volunteers matched for age and sex (for control group) Child and parent/guardian who were willing to participate in the study and provided written informed consent.

-

Exclusion Criteria:Presence of neurological, orthopedic, or psychiatric conditions that could explain the toe walking gait pattern (e.g., cerebral palsy, myopathies, autism spectrum disorders, developmental disorders, neuropathies)

-

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 4 to 12 years diagnosed with bilateral idiopathic toe walking and healthy age-matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Elastography measurements (kPa) of the gastrocnemius muscle and Achilles tendon in children with idiopathic toe walking compared to healthy controls | At study visit (baseline, cross-sectional)
  The gastrocnemius is a biarticular muscle, and its stiffness may be influenced by ankle dorsiflexion and plantarflexion. In the present study, all measurements were performed with the child in the prone position. In children with idiopathic toe walking, both lower extremities were evaluated with the knees extended and the feet hanging off the examination table. Tissue elasticity (kPa) was measured from the medial gastrocnemius and Achilles tendon in three different ankle positions: neutral, passive dorsiflexion, and passive plantarflexion. For each region of interest, five measurements were obtained and averaged.Gastrocnemius muscle and Achilles tendon length was also recorded. For the control group, the same measurements were performed on the dominant lower extremity. The dominant leg was determined by asking the child which foot they would use to kick a ball.

SECONDARY OUTCOMES:
Passive and active ankle dorsiflexion angles measured with a manual goniometer in knee flexion and extension | At study visit (baseline, cross-sectional)
  Bilateral passive and active ankle dorsiflexion angles are measured by using a manual goniometer with the knee positioned in both flexion and extension by the same clinician each time, for both groups
Toe Walking Severity Scale | At study visit (baseline, cross-sectional)
  The Toe Walking Severity Scale is used to evaluate the severity of idiopathic toe walking in children. Parents were asked how often their child walks on toes during the day.
Foot Posture Index | At study visit (baseline, cross-sectional)
  The Foot Posture Index (FPI) was used to evaluate the alignment of the feet and anatomical segments. The FPI, based on the scoring of six different criteria, provided information on whether the foot posture was pronated, neutral, or supinated. The Foot Posture Index scores of children with idiopathic toe walking (ITW) and those in the control group were also compared.
The Pediatric Outcomes Data Collection Instrument | At study visit (baseline, cross-sectional)
  The Pediatric Outcomes Data Collection Instrument (PODCI), a parent-reported questionnaire consisting of 86 items, was used to assess the child's functional status. The two groups were also compared using this instrument.

CONTACTS AND LOCATIONS:
Locations (1):
- Fatih Sultan Mehmet Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided